CLINICAL TRIAL: NCT06845540
Title: Oral Metformin in the Treatment of Melasma: a Prospective Trial in Latin American Women
Brief Title: Oral Metformin for Treating Melasma in Latin American Women
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Puerto Rico (Other)
Responsible Party: Principal Investigator, Cristina Brau-Javier, MD, Associate Professor, University of Puerto Rico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2406248489
Record Dates: First submitted 2025-02-19; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Melasma
Keywords: melasma; metformin
MeSH Terms: conditions — Melanosis | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Metformin (Experimental): Participants received oral metformin tablets, starting at 500 mg once daily. At week 4, those who tolerated the medication increased to 500 mg twice daily for the remainder of the study.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Participants received oral metformin tablets for the treatment of melasma. The initial dose was 500 mg once daily for four weeks. At week 4, participants who tolerated the medication well increased their dose to 500 mg twice daily for the remaining eight weeks of the study. Participants were instructed to avoid other melasma treatments during the trial and to use sunscreen (SPF 30 or higher) daily.

SUMMARY:
The goal of this clinical trial is to learn if metformin can treat melasma in Latin American women. The main question it aims to answer is:

- Can metformin help reduce the dark patches of melasma?

Researchers will test two different doses of metformin (500 mg and 1000 mg) to see if either one helps improve melasma.

Participants will:

* Take a metformin pill every day for three months.
* Go to the clinic twice: once at the beginning and once at the end of the study.
* Get a phone call from the researchers to check how they're doing and ask about any changes or side effects.

ELIGIBILITY:
Inclusion Criteria: Latin American women aged 21 years or older, diagnosed epidermal or mixed melasma

Exclusion Criteria: pregnancy, breastfeeding, use of hydroquinone or tretinoin within 2 months before the study, or undergoing laser treatment, peels, microdermabrasion, or microneedling within 2 months of the study. Patients with a history of renal or liver disease, metformin allergy, diabetes, hypoglycemia, or those on medications that could interact with metformin will also be excluded.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-20 (Estimated); Primary Completion 2025-05-22 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in modified Melasma Area and Severity Index (mMASI) score from baseline to week 12 | Baseline (Week 0) to Week 12
  The primary outcome measure will be the change in melasma severity as assessed by the modified Melasma Area and Severity Index (mMASI) score. The mMASI score will be recorded at baseline (week 0) and at the end of the study (week 12). A blinded investigator will evaluate the participants' melasma severity using this validated scoring system, with a lower mMASI score indicating improvement in melasma.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Brau, Principal Investigator — University of Puerto Rico
Locations (1):
- Administración de Servicios Médicos (ASEM) Clinicas Externas, San Juan, PR, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (mMASI scores, Global Melasma Severity Assessment, and reported adverse events) will be shared with researchers upon request. Data will be available after study completion, pending approval from the principal investigator and institutional review board (IRB). Access will be granted through a secure repository or data-sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: IPD and supporting information will be available starting 6 months after study completion. Data will be accessible for 5 years following publication of the primary study results.
Access Criteria: De-identified individual participant data (mMASI scores, Global Melasma Severity Assessment scores, and reported adverse events) will be shared upon reasonable request. Access will be granted to qualified researchers affiliated with academic or healthcare institutions, subject to approval by the principal investigator and a data-sharing agreement. Requests should be submitted via email to the principal investigator, and approved researchers will receive access through a secure repository.